CLINICAL TRIAL: NCT05622760
Title: Audiovisual Informative Project for the Participants of the Cervical Cancer Screening in Osakidetza
Brief Title: Impact of the Different Information Channels in Reducing Anxiety in Participants of Cervical Cancer Screening
Acronym: DICRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DICRA
Record Dates: First submitted 2022-10-17; First posted 2022-11-21 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Uterine Cervical Neoplasms; Early Detection of Cancer; Anxiety; Clinical Trial
Keywords: uterine cervical neoplasms; anxiety; early detection of cancer; uterine cervical cancer screening; cervical cancer screening; cervical cancer; clinical trial; audiovisual intervention
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Clinical trial on quality of life where there are 2 groups. After signing the informed consents and completing the anxiety surveys, each participant is randomized and given the corresponding envelope.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization code is only known to a collaborator who fills the envelopes according to said code. The envelopes are distributed in order of arrival at the study, the researcher in charge of distributing them and recording the information does not know the randomization code. At the end of the study and registering all the data, the collaborator who has the code will deliver it to the principal investigator of the study.
  In all the envelopes there is some type of information so that the patients are also blind. The experimental group is given a sheet with the links to the videos and the other group is given written information, which is available on the health organization's website. In this way, no group feels that it does not receive information and we control said bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audiovisual information (Experimental): Group of participants to whom the information is given through an audiovisual medium.
  Interventions: Other: Audiovisual information
- Written information (Placebo Comparator): Group of participants to whom the information is given through the writing that is available on the website of the health organization.
  Interventions: Other: Written information

INTERVENTIONS:
Other: Audiovisual information — The information provided to this group is in audiovisual format. This information is what has been designed with the aim of reducing the level of anxiety of patients who participate in cervical cancer screening.
  Arms: Audiovisual information
Other: Written information — The information provided to this group is in written format. This information is what is distributed to patients in the midwife's consultation and is available on the website of the health organization (Osakidetza)
  Arms: Written information

SUMMARY:
When participating in population-based screening for cervical cancer, women experience great anxiety during the weeks of waiting since they learn that they have an altered screening result until the colposcopy is performed. In this study we want to verify how anxiety decreases when the information is improved and an audiovisual support is added when giving it.

DETAILED DESCRIPTION:
This study is designed as a double-blind clinical trial. Candidate patients for this study are women referred to a colposcopy consultation after an altered result of the screening test. Those women who have previously been in the colposcopy consultation or have had this test performed in a private center are excluded.

The initial recruitment is done by telephone. If they accept, they are given an appointment at the hospital one day where, after being informed again and signing the informed consent, they are randomized and assigned a group. There are 2 groups, in one they receive an envelope with the information in writing that was created in Osakidetza and is available on the website of said organization, and the other group receives a sheet with the links to the videos created for this study in the same envelope. In this way, both groups assume that they are receiving information and we avoid bias. The principal investigator is the one who carries out this phase and distributes the envelopes, but is unaware of their contents. Previously, a collaborator fills in the envelopes according to the randomization code and indicates outside the envelope the order in which they should be delivered. Only she knows the randomization code and she will not reveal it until the end of the study.

To analyze the level of anxiety, the participants will fill out 2 scales before receiving the information, and they will return them on the day of the colposcopy before performing it. The scales used are the Spielberger´s State-trait anxiety inventory (STAI) and the Cohen´s PerceivedStress Scale 14 (PSS14). The STAI scale has 40 items, scored from 0 (never) to 3 (very much) points. The final result can range between 0 and 60, higher scores are related to a higher level of anxiety. The PSS14 scale consists of 14 items with a five-point scale response format (0 is never and 4 is very often). The scale scores from 0 to 56; higher scores indicate higher perceived stress.

It will also be analyzed whether the waiting time until the colposcopy and the level of academic studies influence the level of anxiety. And the perception of the colposcopy will be analyzed, with the VAS scale, according to their level of anxiety and the way they received the information.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participate in the Osakidetza cervical cancer screening program and are referred to the colposcopy consultation of the Hospital Universitario Donostia due to an altered screening test.

Exclusion Criteria:

* Patients who have previously been in the colposcopy consultation or have gone to a private center to receive information about their altered result or to undergo colposcopy.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This clinical trial is aimed at all people with a cervix, regardless of the gender that represents them. Although the vast majority are women, men with a cervix can participate.
Enrollment: 140 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Change in the level of anxiety measured by the STAI scale according to the information format | Less than 6 weeks between the call notifying the altered result and the colposcopy
  Change in the level of anxiety according to the information format Compare the level of anxiety between who have the information in audiovisual format and who have the traditional model in written format. For the analysis we will use the STAI (described in Study description).
  The analysis of the results will be done by comparing the basic situation of each participant and the response to the same survey after having the information provided. On the other hand, the results of the surveys between both randomized groups will be compared after having access to the information studied.
Change in the level of anxiety measured by the PSS14 scale according to the information format | Less than 6 weeks between the call notifying the altered result and the colposcopy
  Change in the level of anxiety according to the information format Compare the level of anxiety between who have the information in audiovisual format and who have the traditional model in written format. For the analysis we will use the PSS14 (described in Study description).
  The analysis of the results will be done by comparing the basic situation of each participant and the response to the same survey after having the information provided. On the other hand, the results of the surveys between both randomized groups will be compared after having access to the information studied.

SECONDARY OUTCOMES:
Influence of waiting time for colposcopy on anxiety measured by the STAI scale | 6 weeks maxium
  In this secondary objective, we analyze whether the waiting time from the day the patient knows that she has an altered test until the day of the colposcopy influences the level of anxiety. Generally, the patient has to wait from 2 to 6 weeks from being notified of the altered result until the colposcopy. We are going to group the patients into 3 groups (from 0 to 2 weeks of waiting, from 2 to 4 weeks and from 4 to 6 weeks of waiting) and we will compare the results of the STAI scale to see if this factor is significant in their perception of emotional stress.
Influence of waiting time for colposcopy on anxiety measured by the PSS14 scale | 6 weeks maxium
  In this secondary objective, we analyze whether the waiting time from the day the patient knows that she has an altered test until the day of the colposcopy influences the level of anxiety. Generally, the patient has to wait from 2 to 6 weeks from being notified of the altered result until the colposcopy. We are going to group the patients into 3 groups (from 0 to 2 weeks of waiting, from 2 to 4 weeks and from 4 to 6 weeks of waiting) and we will compare the results of the PSS14 scale to see if this factor is significant in their perception of emotional stress.
Influence of academic level on anxiety measured by the STAI scale | 6 weeks maxium
  The level of anxiety obtained through the STAI scale score will be stratified in the 6 educational level categories (none, primary, secondary, high school, university or professional training) to see if there are significant differences between them.
Influence of academic level on anxiety measured by the PSS14 scale | 6 weeks maxium
  The level of anxiety obtained through the PSS14 scale score will be stratified in the 6 educational level categories (none, primary, secondary, high school, university or professional training) to see if there are significant differences between them.
Change in colposcopy pain perception according to anxiety level measured by the STAI scale | 6 weeks maxium
  We are going to analyze the pain perceived during the colposcopy, using the VAS scale (Visual Analogue Scale of pain) and we will compare them according to the level of anxiety detected in the STAI scale. We want to determine whether the perception of pain worsens at a higher level of anxiety.
Change in colposcopy pain perception according to anxiety level measured by the PSS14 scale | 6 weeks maxium
  We are going to analyze the pain perceived during the colposcopy, using the VAS scale (Visual Analogue Scale of pain) and we will compare them according to the level of anxiety detected in the PSS14 scale. We want to determine whether the perception of pain worsens at a higher level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: David Del Valle, MD, Principal Investigator — Osakidetza
Locations (1):
- Donostia University Hospital, San Sebastián, Guipuzcoa, Spain

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Remor E. Psychometric properties of a European Spanish version of the Perceived Stress Scale (PSS). Span J Psychol. 2006 May;9(1):86-93. doi: 10.1017/s1138741600006004. PMID 16673626